CLINICAL TRIAL: NCT05515601
Title: A Bioequivalence Study of Subcutaneous Injections of Mirikizumab Reference Solution Using an Investigational 1-mL Autoinjector and Mirikizumab Test Solution Formulation Using an Investigational 1-mL Autoinjector in Healthy Participants
Brief Title: A Bioequivalence Study of Mirikizumab (LY3074828) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17327; I6T-MC-AMBT (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-08-24; First posted 2022-08-25 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirikizumab (Reference) (Experimental): 200 milligram (mg) of mirikizumab as reference formulation [100 mg/milliliter (mL)], 2 × 1-mL autoinjector administered as a subcutaneous (SC) injection into the arm/thigh/abdomen on day 1.
  Interventions: Drug: Mirikizumab
- Mirikizumab (Test) (Experimental): 200 mg of mirikizumab as test formulation (100 mg/mL), 2 × 1-mL autoinjector administered as a SC injection into the arm/thigh/abdomen on day 1.
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered SC.

SUMMARY:
The main purpose of this study is to evaluate amount of mirikizumab (test) that gets into the blood stream and how long it takes the body to get rid of it, when given via autoinjector compared to mirikizumab (reference) solution given via autoinjector. The information about any adverse effects experienced will be collected and the tolerability of mirikizumab will also be evaluated.

Screening is required within 35 days prior to enrolment. For each participant, the total duration of the clinical trial will be about 17 weeks including screening.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Have a body mass index( BMI) within the range of 18.0 to 34.0 kg/m2, inclusive.
* are males or non-pregnant women of childbearing potential (WOCBP) or women not of childbearing potential (WNOCBP).

Exclusion Criteria:

* Have significant allergies to humanized monoclonal antibodies or known allergies to mirikizumab, related compounds or any components of the formulation, or history of significant atopy
* Have an abnormal blood pressure, pulse rate, or temperature as determined by the investigator
* Intend to use over-the-counter or prescription medication, including herbal medications and traditional medications, within 7 days prior to dosing
* Are lactating or pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - Altasciences Clinical Los Angeles, Inc, Cypress, California
  - LabCorp CRU, Inc., Daytona Beach, Florida
  - Axis, Dilworth, Minnesota
  - QPS, Springfield, Missouri
  - Labcorp Clinical Research LP, Dallas, Texas
  - LabCorp CRU, Inc., Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otani Y, Feagan BG, D'Haens GR, Escobar R, Morris NJ, Payne CD, Ugolini Lopes M, Zhang X. Pharmacokinetic Comparability and Safety Between Original and Citrate-Free Mirikizumab Formulations for Subcutaneous Injections: Results from Three Clinical Trials. Adv Ther. 2025 May;42(5):2369-2384. doi: 10.1007/s12325-025-03158-y. Epub 2025 Mar 21. PMID 40117091

RESULTS

PARTICIPANT FLOW:
Groups:
- 200 Milligram (mg) Mirikizumab (Reference): Abdomen: Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL (milliliter) autoinjector administered as a subcutaneous (SC) injection into the abdomen on day 1.
- 200 mg Mirikizumab (Reference): Arm: Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL autoinjector administered as a SC injection into the arm on day 1.
- 200 mg Mirikizumab (Reference): Thigh: Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL autoinjector administered as a SC injection into the thigh on day 1.
- 200 mg Mirikizumab (Test): Abdomen: Participants received 200 mg mirikizumab test formulation (100 mg/mL), 2 × 1-mL autoinjector administered as a SC injection into the abdomen on day 1.
- 200 mg Mirikizumab (Test): Arm: Participants received 200 mg mirikizumab test formulation (100 mg/mL), 2 × 1-mL autoinjector administered as a SC injection into the arm on day 1.
- 200 mg Mirikizumab (Test): Thigh: Participants received 200 mg mirikizumab test formulation (100 mg/mL), 2 × 1-mL autoinjector administered as a SC injection into the thigh on day 1.
Period: Overall Study
Arm/Group | 200 Milligram (mg) Mirikizumab (Reference): Abdomen | 200 mg Mirikizumab (Reference): Arm | 200 mg Mirikizumab (Reference): Thigh | 200 mg Mirikizumab (Test): Abdomen | 200 mg Mirikizumab (Test): Arm | 200 mg Mirikizumab (Test): Thigh
Started | 63 | 69 | 67 | 66 | 66 | 65
Received at Least 1 Dose of Study Drug | 63 | 69 | 67 | 66 | 66 | 65
Completed | 62 | 66 | 65 | 65 | 64 | 64
Not Completed | 1 | 3 | 2 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 200 mg Mirikizumab (Reference): Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL autoinjector administered as a SC injection into the arm/thigh/abdomen on day 1.
- 200 mg Mirikizumab (Test): Participants received 200 mg mirikizumab test formulation (100 mg/mL), 2 × 1-mL autoinjector administered as a SC injection into the arm/thigh/abdomen on day 1.
- Total: Total of all reporting groups
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test) | Total
Number analyzed (Participants) | 199 | 197 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (13.0) | 41.1 (12.2) | 40.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 104 | 202
  Male | 101 | 93 | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 33 | 69
  Not Hispanic or Latino | 163 | 164 | 327
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 30 | 59
  White | 150 | 152 | 302
  More than one race | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 199 | 197 | 396

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Mirikizumab
Description: PK: Cmax of mirikizumab was evaluated.
Time Frame: Predose on Day 1, Day 3, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 postdose
Population: All participants who received at least one dose of study drug (mirikizumab) and had evaluable PK data. Participants were excluded from the PK analysis set in the event of 1) a device malfunction, 2) administration of only 1 of the 2 x 1-mL autoinjector doses, or 3) administration of an incorrect or incomplete dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Number analyzed (Participants) | 196 | 192
micrograms per milliliter (μg/mL) | 13.0 (42) | 12.9 (40)
Statistical Analysis 1: Comparison: 200 mg Mirikizumab (Reference) vs 200 mg Mirikizumab (Test); Test type: Other — A linear fixed-effects model is used to estimate the relative bioavailability; Ratio of Geometric least squares mean = 0.986, 90% CI 2-sided [0.929 to 1.05]

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of Mirikizumab
Description: PK: AUC[0-∞] of Mirikizumab was evaluated.
Time Frame: Predose on Day 1, Day 3, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/mL)
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Number analyzed (Participants) | 195 | 192
microgram*day per milliliter (μg*day/mL) | 229 (43) | 232 (42)
Statistical Analysis 1: Comparison: 200 mg Mirikizumab (Reference) vs 200 mg Mirikizumab (Test); Test type: Other — A linear fixed-effects model is used to estimate the relative bioavailability; Ratio of Geometric least squares mean = 1.01, 90% CI 2-sided [0.948 to 1.08]

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC[0-tlast]) of Mirikizumab
Description: PK: AUC[0-tlast] of Mirikizumab was evaluated.
Time Frame: Predose on Day 1, Day 3, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71 and Day 85 postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*day/mL
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Number analyzed (Participants) | 193 | 187
μg*day/mL | 225 (42) | 231 (41)
Statistical Analysis 1: Comparison: 200 mg Mirikizumab (Reference) vs 200 mg Mirikizumab (Test); Test type: Other — A linear fixed-effects model is used to estimate the relative bioavailability; Ratio of Geometric least squares mean = 1.02, 90% CI 2-sided [0.960 to 1.09]

ADVERSE EVENTS:
Time Frame: Baseline Up To 85 Days
Description: All participants who received at least one dose of study drug.
Groups:
- 200 mg Mirikizumab (Reference): Abdomen: Participants received 200 mg mirikizumab reference formulation (100 mg/mL), 2 × 1-mL autoinjector administered as a SC injection into the abdomen on day 1.
Arm/Group | 200 mg Mirikizumab (Reference): Abdomen | 200 mg Mirikizumab (Reference): Arm | 200 mg Mirikizumab (Reference): Thigh | 200 mg Mirikizumab (Test): Abdomen | 200 mg Mirikizumab (Test): Arm | 200 mg Mirikizumab (Test): Thigh
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/69 | 0/67 | 0/66 | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/69 | 0/67 | 0/66 | 0/66 | 0/65
Other Adverse Events (participants affected / at risk) | 11/63 | 12/69 | 13/67 | 7/66 | 11/66 | 12/65
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Mirikizumab (Reference): Abdomen (N=63) | 200 mg Mirikizumab (Reference): Arm (N=69) | 200 mg Mirikizumab (Reference): Thigh (N=67) | 200 mg Mirikizumab (Test): Abdomen (N=66) | 200 mg Mirikizumab (Test): Arm (N=66) | 200 mg Mirikizumab (Test): Thigh (N=65)
Injection site reaction (General disorders) | 10 (19) | 10 (19) | 12 (24) | 4 (7) | 6 (8) | 9 (16)
Headache (Nervous system disorders) | 2 (3) | 4 (4) | 2 (2) | 3 (3) | 7 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT05515601/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT05515601/SAP_001.pdf